CLINICAL TRIAL: NCT00975143
Title: A Double-Blind, Randomized, Phase III, Parallel Group Study Evaluating the Efficacy and Safety of CIP-Isotretinoin in Patients With Severe Recalcitrant Nodular Acne
Brief Title: Efficacy and Safety of CIP-Isotretinoin in Patients With Severe Recalcitrant Nodular Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cipher Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISOCT.08.01
Record Dates: First submitted 2009-09-09; First posted 2009-09-11 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Severe Nodular Acne
Keywords: isotretinoin; dermatology; skin
MeSH Terms: interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CIP-Isotretinoin (Experimental)
  Interventions: Drug: CIP-Isotretinoin
- Isotretinoin (Active Comparator)
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: CIP-Isotretinoin — 0.5 mg/kg/day for 4 weeks, and 1 mg/kg/day for 16 weeks, taken orally, twice daily.
  Arms: CIP-Isotretinoin
Drug: Isotretinoin — 0.5 mg/kg/day for 4 weeks, and 1 mg/kg/day for 16 weeks, taken orally, twice daily.
  Arms: Isotretinoin

SUMMARY:
The purpose of this study is to compare the efficacy and safety of CIP-Isotretinoin and a marketed (generic) formulation of isotretinoin when both are administered twice daily with meals.

ELIGIBILITY:
Inclusion Criteria:

* Severe recalcitrant nodular acne, which in the opinion of the investigator is compatible with isotretinoin treatment.
* Ten (10) or more nodular lesions (facial and/or truncal).
* Treatment-naïve patients without any prior exposure to systemic isotretinoin or other retinoids.
* Age between 12 and 54 years.
* Weight between 40 and 110 kg.
* Negative serum human chorionic gonadotropin (hCG) pregnancy test consistent with a non-pregnant state (females only).
* No significant disease or clinically significant finding in a physical examination.
* No clinically significant abnormal laboratory value.
* No clinically significant abnormal vital sign measurement.
* Patients presenting with stable and controlled diabetes mellitus (Types I and II) may be included in the study. However, patients should not have had a hospitalization for any diabetes related complications in the last 12 months, and must be on stable medication for the preceding 6 months. To be included in the study, the patients should have Hemoglobin-A1c values ≤ 6.5% at screening and in the test done 3 - 4 months previously.
* Patients with previously diagnosed Polycystic Ovarian Syndrome (PCOS) may be included in the study if in the opinion of the investigator they do not have any other clinically significant abnormality (e.g. metabolic syndrome or elevated lipids).

Exclusion Criteria:

* Female patients will be excluded from the study if they:

  * Are pregnant;
  * Are at high risk for becoming pregnant or likely to become pregnant during treatment;
  * Will be breast-feeding or considering breast feeding during the course of the study.
* Known history or presence of any clinically significant unstable medical condition(s) which in the opinion of the investigator could pose a risk for the safety of the patient including any previous history of gastrointestinal disease.
* Patients with any skin disease or other condition that might interfere with the evaluation of recalcitrant nodular acne.
* Patients will be interviewed using the SCID-CT current and lifetime modules for Major Depression, Mania, and Psychosis. Patients with a lifetime history of psychosis will be excluded. Patients with a history of major depressive, manic, hypomanic or mixed episodes will not be excluded unless they have had an episode during the preceding year.
* Patients with any past or current psychotic symptoms.
* Patients reporting any suicidal behaviour (including attempts, interrupted attempts, aborted attempts, or other preparatory behaviours), within the past year, or serious suicidal ideation in the past year, will be excluded from study participation.
* A lifetime history of wishing to be dead, non-specific active suicidal thoughts or active suicidal ideation without intent to act will not result in exclusion.
* Known history or suspected carcinoma.
* Known history of liver or kidney disorders (hepatic and renal insufficiency).
* Known history or current pseudotumor cerebri (benign intracranial hypertension).
* Patients with HLA-B27 related disease, rheumatoid arthritis, rickets or other vitamin D depletion disease or phosphate metabolic disease, severe scoliosis > 15 Cobb angle, history of back surgery/injuries, ongoing use of anticonvulsants known to affect bone metabolism and other genetic or acquired rheumatologic and joint diseases.
* All pediatric patients with serum 25-hydroxyvitamin D levels < 20 ng/mL.
* Patients with hearing disorders who in the opinion of the investigator would not be able to participate in audiometric testing for the study.
* Hypersensitivity or idiosyncratic reaction to isotretinoin, Vitamin A and/or any other drug substances with similar activity.
* Allergy to soy beans, soy bean oil or any other ingredients in the study medications.
* On a special diet within four weeks prior to drug administration (e.g., liquid, protein, raw food diet).
* Difficulty consuming two (2) meals a day to sustain weight and health.

Ages: 12 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 925 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J. Leyden, MD, Study Chair — University of Pennsylvania; Guy Webster, MD, Study Chair — Jefferson Medical College of Thomas Jefferson University; Jason A. Gross, PharmD, Study Director — Cipher Pharmaceuticals Inc.
Locations (49):
- United States (37):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Center for Dermatology Clinical Research, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists, Oceanside, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Horizons Clinical Research Center, Denver, Colorado
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - Ameriderm Research, Jacksonville, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Peachtree Dermatology Associates, PC, Atlanta, Georgia
  - MedaPhase Inc., Newnan, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Northwest Clinical Trials, Nampa, Idaho
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - The South Bend Clinic, LLP, South Bend, Indiana
  - Dermatology and Skin Cancer Specialists / Pediaresearch, LLC, Owensboro, Kentucky
  - ActivMed Practices & Research, Haverhill, Massachusetts
  - Great Lakes Research Group, Bay City, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Haber Dermatology, Clinical Research Center, South Euclid, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Paddington Testing Company Inc., Philadelphia, Pennsylvania
  - Radiant Research, Inc., Greer, South Carolina
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Suzanne Bruce and Associates - The Center for Skin Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Stephen Miller, MD, PA Dermatology, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Premier Clinical Research, Spokane, Washington
- Canada (12):
  - Derm Research @ 888 Inc., Vancouver, British Columbia
  - Dermadvances Research, Winnipeg, Manitoba
  - Durondel C.P. Inc, Moncton, New Brunswick
  - Newlab Clinical Research Inc., St. John's, Newfoundland and Labrador
  - UltraNova Skincare, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Windsor Clinical Research, Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at 49 investigational centers in the United States and Canada. Of the 1265 patients screened for the study, a total of 925 were randomized to CIP-Isotretinoin (N=464) or generic Isotretinoin (N=461) between October 2009 and October 2010. Randomization was stratified by gender and study site.
Pre-assignment Details: Reasons for screen failure: patient's decision (83 pts), low disease severity (61), entry criteria (51), psychological disqualification (44), lost to follow-up (33) and low vitamin D levels (33). Washouts were specified for: systemic corticosteroids, spironolactone (30 d), other acne treatment, phenytoin (14 d), topical corticosteroids (7 d).
Groups:
- CIP-Isotretinoin: CIP-Isotretinoin 10 mg and 20 mg capsules taken with meals, at an initial titration dose of approximately 0.5 mg/kg/day, divided into 2 doses for the first 4 weeks, followed by approximately 1 mg/kg/day divided into 2 doses for 16 weeks
- Isotretinoin: (Generic) Isotretinoin 10 mg and 20 mg capsules taken with meals, at an initial titration dose of approximately 0.5 mg/kg/day, divided into 2 doses for the first 4 weeks, followed by approximately 1 mg/kg/day divided into 2 doses for 16 weeks
Period: Overall Study
Arm/Group | CIP-Isotretinoin | Isotretinoin
Started | 464 | 461
Completed Treatment (Week 20) | 403 | 410
Completed | 394 | 401
Not Completed | 70 | 60
Not completed — Adverse Event | 19 | 15
Not completed — Withdrawal by Subject | 15 | 15
Not completed — Lost to Follow-up | 20 | 16
Not completed — Non-compliance | 5 | 8
Not completed — Physician Decision | 1 | 2
Not completed — Details not available | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CIP-Isotretinoin | Isotretinoin | Total
Number analyzed (Participants) | 464 | 461 | 925
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 205 | 192 | 397
  Between 18 and 65 years | 259 | 269 | 528
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (7.5) | 20.7 (6.8) | 20.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 178 | 365
  Male | 277 | 283 | 560
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was designated as Hispanic or Non-Hispanic.
  Participants
    Hispanic or Latino | 59 | 63 | 122
    Not Hispanic or Latino | 405 | 398 | 803
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 380 | 373 | 753
  Canada | 84 | 88 | 172
Nodular Lesion Count [Mean (Standard Deviation); unit: Lesions] — Qualified medical practitioners, blinded to treatment group assignment made counts of nodules in the facial and truncal area. Where possible, the same individual performed all evaluations for a patient.
  Lesions | 18.4 (14.7) | 17.7 (10.8) | 18.0 (12.9)
Inflammatory Lesion Count [Mean (Standard Deviation); unit: Lesions] — Qualified medical practitioners, blinded to treatment group assignment made counts of inflammatory lesions (papules and pustules) in the facial and truncal area. Where possible, the same individual performed all evaluations for a patient.
  Lesions | 37.8 (31.3) | 38.4 (34.5) | 38.1 (33.0)
Physician's Global Severity Assessment (PGSA) [Number; unit: participants] — Acne severity status was graded by the investigator on a 6-point scale, from 0 = Clear (No nodules, pustules or papules visible) to 5 = Very Severe (Highly inflammatory acne covering the affected area, with many nodules and cysts present ). The PGSA was applied to facial lesions only (ie, not conducted on patients with only truncal lesions).
  participants
    1 (Almost clear) | 3 | 2 | 5
    2 (Mild) | 11 | 10 | 21
    3 (Moderate) | 49 | 60 | 109
    4 (Severe) | 329 | 322 | 651
    5 (Very Severe) | 64 | 63 | 127
    Not assessed | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Outcome 1: Change From Baseline in Total Nodular Lesion Count (Facial and Truncal)
Description: The change from Baseline to Week 20 in the total number of nodular lesions was calculated as the Week 20 lesion count minus Baseline lesion count and compared using Analysis of Covariance (ANCOVA), controlling for Baseline total nodular lesion count, gender and analysis site.
  The 95% CI of the adjusted least square mean difference (CIP-ISOTRETINOIN minus Isotretinoin) was also calculated using the ANCOVA model.
  Pre-defined criterion for non-inferiority: upper bound of the 95% CI for the treatment difference < 4.
Time Frame: 20 weeks
Population: Analysis based on the Per Protocol (PP) Population, defined as all randomized patients who were at least 75% compliant with their assigned treatment, had no major study protocol violations, had a Week 20 count of total nodular lesions, and did not use any disallowed medications during the 20 study weeks.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | CIP-Isotretinoin | Isotretinoin
Number analyzed (Participants) | 363 | 361
Lesions | -17.01 (14.26) [-0.2712 to 0.5475] | -16.52 (10.57) [-1.1337 to 3.5338]
Statistical Analysis 1: Comparison: CIP-Isotretinoin vs Isotretinoin; Change from Baseline was calculated as the post-Baseline value minus the Baseline value; Test type: Non-Inferiority or Equivalence — Pre-defined criterion for non-inferiority: upper bound of the 95% CI for the treatment difference < 4; p = 0.5077, ANCOVA — P values are from analysis of covariance (ANCOVA) controlling for Baseline total nodular lesion count, gender and analysis site; The 95% CI of the adjusted least square mean difference (CIP-ISOTRETINOIN minus Isotretinoin) was calculated using the ANCOVA model; LS Mean Difference = 0.1382, 95% CI 2-sided [-0.2712 to 0.5475]

2. Secondary Outcome: Proportion of Patients Who Are Rated as Clear/Almost Clear on the Six-point Physicians' Global Assessment Scale (PGSA).
Description: PGSA categories: 1 (Almost clear); 2 (Mild); 3 (Moderate); 4 (Severe); 5 (Very severe). A grade of either 0 (clear) or 1 (almost clear) on the 6-point PGSA scale within the Week 20 analysis window was considered a success.
Time Frame: 20 weeks
Population: Analysis based on the Per Protocol (PP) Population. Patients with a Baseline PGSA score of 0 or 1 (i.e., who had primarily truncal lesions at Baseline) were excluded from the analysis, as PGSA evaluated facial lesions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CIP-Isotretinoin | Isotretinoin
Number analyzed (Participants) | 348 | 349
percentage of participants | 85.9 [82.3 to 89.6] | 89.4 [86.2 to 92.6]
Statistical Analysis 1: Comparison: CIP-Isotretinoin vs Isotretinoin; The analysis of the secondary efficacy endpoint was based on observed cases only, with no imputation for missing values; Test type: Non-Inferiority or Equivalence — If the two co-primary endpoints were significant, a 95% 2 sided CI on the difference between treatments (CIP-Isotretinoin minus Isotretinoin) was calculated; p > 0.05, Normal approximation; 95% CI on difference in proportions (CIP-Isotretinoin minus Isotretinoin) was estimated using normal approximation; Proportion difference = -3.48, 95% CI 2-sided [-8.4 to 1.4]

3. Primary Outcome: Co-Primary Outcome 2: Proportion of Patients Who Achieve at Least a 90% Reduction in Total Number of Nodular Lesions (Facial and Truncal).
Description: The percentage of patients in each group who achieved ≥90% reduction in the total nodular lesion count from Baseline to Week 20 was calculated along with its 95% CI (normal approximation). A 95% 2-sided CI on the difference between treatments (CIP-ISOTRETINOIN minus Isotretinoin) was also computed.
  Pre-defined criterion for non-inferiority: lower bound of the 95% CI for the treatment difference > -10.
Time Frame: 20 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CIP-Isotretinoin | Isotretinoin
Number analyzed (Participants) | 363 | 361
percentage of participants | 78.8 [74.6 to 83.0] | 80.9 [76.8 to 84.9]
Statistical Analysis 1: Comparison: CIP-Isotretinoin vs Isotretinoin; Test type: Non-Inferiority or Equivalence — Pre-defined criterion for non-inferiority: lower bound of the 95% CI for the treatment difference > -10; p > 0.05, Normal approximation; Proportion difference = -2.10, 95% CI 2-sided [-7.94 to 3.74]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the beginning of double-blind treatment until 30 days after the last study treatment (Week 24). AEs occurring before starting study treatment but after signing the informed consent form were recorded under Medical History.
Description: Adverse events were analyzed based on the Safety Population (defined as all randomized patients who consumed at least one dose of study medication, including those for whom dosing information was unknown), based on the actual treatment received. The Safety Population included 924 patients (CIP-Isotretinoin 464, Isotretinoin 460).
Arm/Group | CIP-Isotretinoin | Isotretinoin
Serious Adverse Events (participants affected / at risk) | 7/464 | 5/460
Other Adverse Events (participants affected / at risk) | 428/464 | 413/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIP-Isotretinoin (N=464) | Isotretinoin (N=460)
Abdominal pain (Gastrointestinal disorders) | 1 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CIP-Isotretinoin (N=464) | Isotretinoin (N=460)
Lip dry (Gastrointestinal disorders) | 209 | 210
Dry skin (Skin and subcutaneous tissue disorders) | 205 | 206
Back pain (Musculoskeletal and connective tissue disorders) | 96 | 89
Dry eye (Eye disorders) | 87 | 78
Arthralgia (Musculoskeletal and connective tissue disorders) | 64 | 60
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 54 | 42
Headache (Nervous system disorders) | 37 | 36
Nasopharyngitis (Infections and infestations) | 36 | 48
Chapped lips (Gastrointestinal disorders) | 34 | 32
Dermatitis (Skin and subcutaneous tissue disorders) | 28 | 23
Blood creatine kinase increased (Investigations) | 26 | 27
Cheilitis (Gastrointestinal disorders) | 26 | 19
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 25 | 16
Upper respiratory tract infection (Infections and infestations) | 25 | 14
Visual acuity reduced (Eye disorders) | 23 | 25

LIMITATIONS AND CAVEATS:
Generic isotretinoin control because Accutane® was discontinued in the US. 201 PPP exclusions (CIP-Isotretinoin 101, Isotretinoin 100) due to discontinuation < Week 20 (61+51), non-compliance with treatment (76+75) or other requirements (≥1 reason).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less